CLINICAL TRIAL: NCT06968832
Title: Project COMET: Hybrid Effectiveness-Implementation Trial of Massed PTSD Treatment in a Community Substance Use Program
Brief Title: Project COMET: Massed Prolonged Exposure for PTSD and SUD
Acronym: PROJECT COMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, San Diego (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Denise Aimee Hien, Helen E. Chaney Endowed Chair in Alcohol Studies; Distinguished Professor, Graduate School of Applied and Professional Psychology, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2024002340; 1R01MH132720-01A1 (NIH)
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Substance Use Disorders (SUD); Comorbidity; Trauma and Stressor Related Disorders
Keywords: Posttraumatic Stress Disorder (PTSD); Substance Use Disorder (SUD); PTSD/SUD Comorbidity; Prolonged Exposure Therapy (PE); Massed Prolonged Exposure (M-PE); Randomized Clinical Trial (RCT); Treatment as Usual (TAU); Integrated PTSD and SUD Treatment; Implementation Science; Trauma-Focused Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Trauma and Stressor Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group randomized controlled trial. Participants will be randomly assigned to receive either (1) Massed Prolonged Exposure (M-PE) therapy integrated within Intensive Outpatient (IOP) Substance Use Disorder (SUD) treatment or (2) Treatment as Usual (TAU) in IOP SUD care, which includes a weekly trauma skills group. The goal is to evaluate the effectiveness of M-PE in improving PTSD and substance use outcomes compared to standard IOP programming.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massed Prolonged Exposure (M-PE) + Intensive Outpatient Program (IOP) (Experimental): Participants randomized to this arm will receive Massed Prolonged Exposure (M-PE) therapy, a gold-standard treatment for PTSD delivered multiple times per week over 2-4 weeks. M-PE will be integrated into the standard Intensive Outpatient Program (IOP) for substance use disorder (SUD) at Gateway Community Services, Inc. This arm is designed to evaluate the effectiveness of delivering M-PE concurrently with SUD treatment in improving PTSD symptoms, reducing substance use, and improving patient-centered outcomes.
  Interventions: Behavioral: Massed Prolonged Exposure Therapy (M-PE)
- Trauma Treatment as Usual (TAU) - IOP with Trauma Skills Group (Active Comparator): Participants randomized to this arm will receive the standard Intensive Outpatient Program (IOP) for substance use disorder (SUD), which includes a weekly trauma skills group as part of usual care. This comparator arm allows for evaluation of whether M-PE enhances outcomes beyond those achieved through trauma-informed IOP care.
  Interventions: Behavioral: Standard outpatient SUD care

INTERVENTIONS:
Behavioral: Massed Prolonged Exposure Therapy (M-PE) — Massed Prolonged Exposure (M-PE) is a trauma-focused, evidence-based behavioral intervention for posttraumatic stress disorder (PTSD). It is delivered over a compressed timeline (e.g., 10 sessions over 2-4 weeks) as opposed to weekly sessions over 3-4 months. This format has been shown to accelerate PTSD symptom reduction and reduce treatment dropout. In this study, M-PE will be delivered concurrently with an Intensive Outpatient Program (IOP) for substance use disorder (SUD) at Gateway Community Services. Sessions will be led by trained clinicians using a standardized PE protocol, with treatment including imaginal exposure, in vivo exposure, and processing.
  Other Names: M-PE
  Arms: Massed Prolonged Exposure (M-PE) + Intensive Outpatient Program (IOP)
Behavioral: Standard outpatient SUD care — Patients randomized to usual care will receive standard intensive outpatient SUD treatment.
  * Resilience group (weekly)
  * Peer support
  * Individual therapy from a variety of modalities
  Other Names: Usual Care Condition
  Arms: Trauma Treatment as Usual (TAU) - IOP with Trauma Skills Group

SUMMARY:
The goal of this clinical trial is to learn if Massed Prolonged Exposure Therapy (M-PE) can improve PTSD symptoms and reduce substance use in adults receiving intensive outpatient (IOP) treatment for substance use disorder (SUD). The main questions it aims to answer are:

* Does M-PE reduce PTSD symptoms more effectively than trauma treatment as usual (TAU)?
* Does M-PE reduce the number of days participants use substances?
* How do patient-centered outcomes (such as depression, suicidal thoughts, and quality of life) differ between M-PE and trauma TAU?
* Researchers will compare M-PE to treatment as usual to see if M-PE leads to better mental health and substance use outcomes and lower dropout rates.

Participants will:

* Attend multiple therapy sessions per week (M-PE) or receive usual care
* Complete assessments at baseline, during treatment, end-of-treatment, 1-month, 3-month, and 6-month follow-up
* Share feedback through surveys and interviews about their experience in the program

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) and substance use disorder (SUD) often co-occur. PTSD+SUD comorbidity is associated with more severe PTSD, worse treatment outcomes for substance use, greater suicide risk and worse functioning than having one of these disorders. First-line treatments for PTSD, particularly Prolonged Exposure Therapy (PE), are effective in treating PTSD among those with a SUD. While PE is one of the most effective treatment options for PTSD among those with PTSD+SUD, effects are smaller and dropout is higher than among people with PTSD without a SUD. A promising way to enhance outcomes is to offer PE in a massed format (M-PE; i.e., multiple sessions per week instead of once weekly).

M-PE has been shown to be effective in improving PTSD symptoms and substantially reducing dropout in outpatient care. Preliminary findings suggest M-PE delivered concurrent to intensive SUD programming is a promising strategy that warrants further study. Evaluating the effectiveness of M-PE delivery in of SUD IOP program in improving PTSD and other mental health outcomes is the necessary next step in this critical research.

The mixed-method two-group Hybrid Type I effectiveness-implementation randomized clinical trial (RCT) aims to determine the effectiveness of M-PE delivery in SUD IOP in reducing dropout rates and improving outcomes as compared to trauma treatment as usual (TAU).

The specific aims are to 1) Compare the effectiveness of M-PE to trauma TAU in IOP SUD treatment in impacting PTSD symptoms and Percent days use of primary substance; 2) Explore differences in treatment arms on patient-centered outcomes, including: a) days use of other (non-primary) substances, b) depressive symptoms, c) functioning, c) quality of life (QoL), e) suicidal ideation, and f) participant satisfaction; 3) Examine gender as a moderator and changes in trauma-related cognitions, cravings, and their temporal association as mediators of change in PTSD and substance use; and 4) Conduct a mixed-method process evaluation to understand patients', providers', and clinical stakeholders' experiences with M-PE, explore barriers and facilitators to integrating M-PE into IOP SUD treatment, and identify strategies for widespread implementation.

Participants will include 168 male and female patients with any trauma type who are participating in IOP SUD program at Gateway Community Services, Inc. Assessments will occur at baseline, and will continue for the duration of treatment, at end-of-treatment, 1-month posttreatment, 3-months posttreatment, and 6-months posttreatment. We will conduct a mixed-method, multi-stakeholder process evaluation with patients, providers, and clinical leaders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Enrolled in SUD treatment at Gateway Community Services
* Meet DSM-5 criteria for a SUD (Tobacco Use Disorder alone not sufficient for inclusion)
* Meet DSM-5 criteria for PTSD
* Able to give informed consent

Exclusion Criteria:

* severe cognitive impairment
* current suicidal or homicidal intent requiring immediate treatment
* current unstable psychotic or manic symptoms not attributable to SUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline; End of Treatment (6 weeks post-randomization); 1-month (10 weeks), 3-month (18 weeks), and 6-month (30 weeks) post-randomization follow-up
  Measures PTSD symptom severity, score range 0-80, higher scores mean greater symptom severity
Time Line Follow back (TLFB) | Baseline; End of Treatment (6 weeks post-randomization); 1-month (10 weeks), 3-month (18 weeks), and 6-month (30 weeks) post-randomization follow-up
  Measures percent days of alcohol or other drug use, score range 0-100%, higher scores indicate greater percent days of use

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline; End of Treatment (6 weeks post-randomization); 1-month (10 weeks), 3-month (18 weeks), and 6-month (30 weeks) post-randomization follow-up
  Depression symptom severity, range = 0-27, higher scores mean greater depression symptom severity
Brief Psychosocial Functioning Inventory (B-IPF) | Baseline; End of Treatment (6 weeks post-randomization); 1-month (10 weeks), 3-month (18 weeks), and 6-month (30 weeks) post-randomization follow-up
  Measures severity of impairment in psychosocial functioning, scores = 0-100, higher scores indicate greater impairment
Brief Substance Craving Scale (BSCS) | Baseline; End of Treatment (6 weeks post-randomization); 1-month (10 weeks), 3-month (18 weeks), and 6-month (30 weeks) post-randomization follow-up
  Assesses craving severity for a primary and, if applicable, secondary substance over the past 24 hours. Includes items on intensity, frequency, duration, and number of craving episodes. Higher scores reflect greater craving.

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Norman Professor Of Clinical, Psychiatry, Ph.D, Principal Investigator — University of California, San Diego
Locations (1):
- Gateway Community Services, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data (IPD) that underlie the results reported in the study, following de-identification and in compliance with IRB and data use agreements. A data dictionary will also be provided to allow for accurate interpretation of variables and data structure. Data will be made available to qualified researchers upon request, following approval of a data use agreement and verification of appropriate data security measures.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The IPD and supporting information will be available beginning 6 months after publication of the primary outcomes and will remain available for 5 years.
Access Criteria: Qualified researchers affiliated with academic institutions or research organizations will be able to request access to the de-identified individual participant data (IPD) and accompanying materials, including the data dictionary and study protocol. Access will include data related to primary and secondary outcomes, as well as adverse events, once appropriate data use agreements are in place.
  Requests must be submitted to the study team and will be reviewed for scientific merit, ethical use, and compliance with institutional and regulatory guidelines. Approved users will be granted access through a secure data-sharing platform or via direct encrypted transfer, in accordance with Rutgers University and sponsor policies on data security and privacy.